CLINICAL TRIAL: NCT07021339
Title: Randomized, Controlled Trial of Anterior Temporal Lobectomy Versus Gross Total Resection in Newly-diagnosed Temporal Glioblastoma (ATLAS/NOA-29)
Brief Title: Anterior Temporal Lobectomy in Temporal Glioblastoma
Acronym: ATLAS/NOA-29
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: University Hospital RWTH Aachen, Department of Neurosurgery (Unknown); Kantonsspital Aarau, Department of Neurosurgery (Unknown); University Hospital Bonn, Department of Neurosurgery (Unknown); Dortmund Hospital, Neurosurgical Department (Unknown); Helios Kliniken, Erfurt, Department of Neurosurgery (Unknown); University Hospital Essen, Department of Neurosurgery and Spine Surgery (Unknown); University Hospital Frankfurt, Department of Neurosurgery (Unknown); University Hospital Giessen, Department of Neurosurgery (Unknown); University Medical Center Göttingen, Department of Neurosurgery (Unknown); University Medical Center Hamburg-Eppendorf, Department of Neurosurgery (Unknown); Heidelberg University Hospital, Department of Neurosurgery (Unknown); Jena University Hospital, Department of Neurosurgery (Unknown); University of Cologne, Center of Neurosurgery Department of General Neurosurgery (Unknown); University Hospital Leipzig, Department of Neurosurgery (Unknown); University Medical Center Schleswig-Holstein/Lübeck, Department of Neurosurgery (Unknown); Medical Faculty University Hospital Magdeburg, University Clinic for Neurosurgery (Unknown); University Medical Center Mainz, Department of Neurosurgery (Unknown); University Hospital Mannheim, Medical Faculty Mannheim, Department of Neurosurgery (Unknown); Klinikum Rechts der Isar, Technical University of Munich, Department of Neurosurgery (Unknown); LMU University Hospital, Department of Neurosurgery (Unknown); University Hospital of Münster, Department of Neurosurgery (Unknown); University Hospital Regensburg, Department of Neurosurgery (Unknown); University Medical Centre Rostock, Department of Neurosurgery (Unknown); University Hospital Tübingen, Department of Neurosurgery (Unknown); University Hospital Ulm/Günzburg, University of Ulm, Department of Neurosurgery (Unknown); Medical University of Vienna, Department of Neurosurgery (Unknown)
Responsible Party: Principal Investigator, Matthias Schneider, PD Dr. med., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70114652; 290/23 (Other: University Hospital Bonn, Department of Neurosurgery)
Record Dates: First submitted 2025-03-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Newly-diagnosed Glioblastoma; Temporal Lobe
Keywords: ATLAS/NOA-29; ATLAS; NOA-29; Anterior temporal lobectomy; gross total resection
MeSH Terms: interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gross total resection (GTR) (Active Comparator): Complete resection of the contrast-enhancing tumor in Magnetic Resonance Imaging (MRI)
  Interventions: Procedure: Gross Total Resection (GTR)
- Anterior temporal lobectomy (ATL) (Experimental): Anterior temporal lobectomy
  Interventions: Procedure: Anterior temporal lobectomy (ATL)

INTERVENTIONS:
Procedure: Anterior temporal lobectomy (ATL) — Patients assigned to the experimental group will undergo an anterior temporal lobectomy (ATL) according to established protocols adapted from epilepsy surgery. ATL is a reproducible and anatomically well-defined procedure routinely performed in patients with pharmacoresistant temporal lobe epilepsy. On the non-dominant hemisphere, the neocortical resection typically extends 6.5 cm posteriorly from the temporal pole, while on the dominant side, the resection length is limited to 4.0 cm, both measured along the superior temporal gyrus and guided by the Sylvian fissure. Language dominance is determined based on handedness, as specified in the inclusion criteria. In most cases, the lateral neocortical segment can be removed en bloc.
  The mesial component of ATL encompasses resection of the uncus, amygdala, and the anterior hippocampus, typically including both the head and body. Resection is carried out to the level of the tectal plate or, at minimum, to the lateral mesencephalic sulcus.
  Arms: Anterior temporal lobectomy (ATL)
Procedure: Gross Total Resection (GTR) — Patients will be surgically treated with GTR in terms of removing 100% of the tumor tissue in gadolinium-enhanced MRI.
  Arms: Gross total resection (GTR)

SUMMARY:
The ATLAS/NOA-29 trial is a prospective, multicenter, phase III randomized controlled study evaluating whether anterior temporal lobectomy (ATL), a standardized resection technique adapted from epilepsy surgery, improves clinical outcomes in patients with newly diagnosed glioblastoma of the anterior temporal lobe compared to conventional gross-total resection (GTR). The rationale is based on the concept of glioblastoma as a diffusely connected tumor network, with infiltrative spread extending beyond MRI-detectable tumor margins. ATL offers a reproducible supramarginal resection approach within anatomical boundaries that are routinely respected in epilepsy surgery.

Patients are randomized intraoperatively in a 1:1 ratio following histopathological confirmation via intraoperative frozen section procedure. The trial's primary objective is to demonstrate superiority of ATL in overall survival (OS), while confirming non-inferiority in health-related quality of life (QoL), measured by the global health status scale of the European Organisation for Research and Treatment of Cancer (EORTC) - Quality of Life Questionnaire Core 30 (QLQ-C30). Secondary outcomes include progression-free survival (PFS), seizure control, neurocognitive functioning, and longitudinal assessments of selected EORTC QLQ-C30 and BN20 domains. A total of 178 patients will be enrolled over three years, with a minimum follow-up of three years. An interim safety analysis after inclusion of 57 patients will assess functional outcome differences using the modified Rankin Scale (mRS) at 6 months postoperatively. The study is powered (>80%) to detect a survival benefit assuming a median OS increase from 17 to 27.5 months. If proven superior to GTR, ATL could emerge as the preferred surgical strategy for isolated temporal lobe glioblastoma, offering robust evidence in favor of extending supramarginal resection principles to the broader context of glioblastoma care.

ELIGIBILITY:
* Suspected glioblastoma with contrast-enhancement in preoperative MRI
* Diffuse high-grade glioma in frozen section procedure, newly-diagnosed
* Tumor localization (in gadolinium-enhanced MRI): solely temporal, non-dominant side (right hemisphere in right-handed patients, or left-handed patients after testing for dominance): within 6.5 cm from the temporal pole; dominant side (left hemisphere in right-handed patients, all left-handed patients unless additional testing for dominance performed): within 4.0 cm from the temporal pole, as determined dorsally along the Sylvian fissure.
* Macroscopic complete resection (no remaining contrast-enhancing tumoral lesion on early postoperative MRI) is achievable (decision of the treating neurosurgeon)
* In case further T1-contrast-enhancing and/or T2/FLAIR lesions are detected beyond the resection margins (6.5 cm on the non-dominant side and 4.0 cm on the dominant side), these lesions are not attributed to the tumor (except perifocal edema) but to other conditions according to the local treating neurosurgeon
* ≥ 18 and < 75 years of age
* KPS ≥ 70%
* Estimated life expectancy of at least 6 months
* Written informed consent
* Cognitive state to understand the rationale and necessity of the study therapy and procedures
* Patient compliance and geographic proximity that allow adequate follow-up
* For patients with childbearing potential: negative serum pregnancy test (beta-HCG) at baseline visit, patient's commitment to use an approved contraceptive method during the trial and for 3 months after (Pearl index < 1%)
* Adequate organ function at baseline visit that does not preclude alkylating chemotherapy and neurosurgical procedures (all criteria required):

  * Adequate bone marrow reserve: white blood cell (WBC) count ≥ 3.000/µl; granulocyte count > 1.500/µl; platelets ≥ 100.000/µl; haemoglobin ≥ 10 g/dl
  * Adequate liver function: bilirubin < 1.5 times above upper limit of normal range (ULN); alanine transaminase (ALT/SGPT) and aspartate transaminase (AST/ALAT) < 3 times ULN
  * Adequate renal function: creatinine < 1.5 times ULN
* Adequate blood clotting: Partial Thromboplastin Time (PTT) not exceeding the upper limit of normal range and International Normalized Ratio (INR) <1.5; in case of intake of anticoagulant medication or platelet function inhibitors, the coagulation analysis must show no detectable effect in specific blood tests (as described below) at the time of surgery, and discontinuation of the anticoagulant medication must be justifiable for at least 1 week postoperatively

  * Direct acting oral anticoagulants (e.g., rivaroxaban, apixaban, edoxaban, dabigatran): anti-Factor Xa (aFXa)-activity within the normal range (rivaroxaban, apixaban, edoxaban), TT/TCT (thrombin clotting time) or ecarin clotting time (ECT) not exceeding the upper limit of normal range (Dabigatran) or verification of subtherapeutic drug levels (apixaban, edoxaban, rivaroxaban, dabigatran)
  * Vitamin K antagonists (coumarins): INR < 1.5
  * Unfractionated heparin (UFH) and argatroban: activated Partial Thromboplastin Time (aPTT) not exceeding the upper limit of normal range
  * Fractionated heparin/low-molecular-weight heparin (e.g., dalteparin, enoxaparin), heparinoid (e.g., fondaparinux, danaparoid): aFXa-activity within the normal range
  * Antiplatelet agents (aspirin, clopidogrel, prasugrel, ticagrelor): platelet function analyzer (PFA) test not exceeding the upper limit of normal range (aspirin), whole blood aggregometry not below lower limits of normal range (clopidogrel, prasugrel, ticagrelor)

For details see study protocol.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From randomization until death or 36 months after recruitment of the last patient
  OS in the modified intention to treat (mITT) population of patients with glioblastoma, Central Nervous System (CNS) World Health Organization (WHO) grade 4, Isocitrate Dehydrogenase wild-type (IDHwt)
Patient-reported Quality of Life | From randomization until death or 36 months after recruitment of the last patient
  In case of significant OS differences, the patient-reported QoL domain "global health status" (EORTC QLQ-C30 questionnaire) in the modified intention to treat (mITT) population is the co-primary endpoint. Over-all superiority of ATL requires significantly prolonged OS and non-inferiority regarding the development of the global health status over time in the mITT population.

SECONDARY OUTCOMES:
Progression-free survival | PFS is measured from randomization at the day of surgery until progression or death. PFS will be assessed at the 12-week follow-up visit and at all subsequent visits scheduled at 12-week intervals up to three years.
  Progression is defined as the first documented evidence of progression of disease according to the Response Assessment in Neuro-Oncology 2.0 (RANO 2.0) criteria. Progression will be evaluated using the RANO (Response Assessment in Neuro-Oncology) 2.0. criteria.
Neurocognitive Outcome | Cognitive performance across all domains will be quantitatively assessed at baseline (preoperatively), and at follow-up visits on day 90 (visit 8) and one year after surgery (visit 11).
  All patients will undergo testing with the Brain Lesion Tracking Test (BLTT). The test covers all relevant domains of neurocognition-including episodic and semantic memory as well as executive functions-without excluding patients due to neurological impairments such as visual deficits or hemiparesis.
  The BLTT includes interlocking word list learning with delayed free recall and recognition, semantic word generation and fluency, phonemic fluency, reverse digit span, and incidental memory, providing a rapid screening of neurocognitive function. Results are categorized into three performance domains: executive functions, episodic memory, and semantic memory. In addition, figural memory is assessed through a visual recognition task involving drawn objects presented on a series of cards.
Karnofsky Performance Scale | KPS will be assessed at baseline, on postoperative day 1, and at follow-up visits on days 3, 14, 30, and 90, and subsequently at 12-week intervals.
  Karnofsky Performance Scale (KPS) is an attempt to quantify cancer patients' general well-being and activities of daily life. The KPS ranking runs from 100 to 0, where 100 is "perfect" health and 0 is death.
Seizure outcome | Seizure outcome will be assessed at the 12 weeks, the 6 months and all 12 week follow-up examination.
  Analysis of postoperative seizure outcome will be assessed referring to the ILAE classification system in the course of epilepsy surgical procedures: seizure freedom (ILAE class 1) will be de-fined as a favorable seizure outcome; ILAE classes 2-6 (i.e. pure auras, rare to no improvement and worsening of seizure frequency) will be referred to as unfavorable seizure outcome.
Modified Rankin Scale assessment (mRS) | The mRS will be assessed at baseline, on postoperative day 1, and at follow-up visits on days 3, 14, 30, and 90, and subsequently at 12-week intervals.
  The mRS will be used for measuring the degree of disability or dependence in the daily activities of patients. The mRS ranking runs from 0 to 6, where 0 is "perfect" health and 6 is death. Furthermore, 6 months after randomization of the 57th patient there will be carried out an interim safety analysis, which will evaluate differences in clinical performance (mRS) between the experimental and conventional intervention groups.
Quality-of-life (QoL) | QoL will be assessed at baseline, at follow-up visits on days 14, 30, and 90, and subsequently at 24-week intervals.
  The EORTC quality of life (QoL) questionnaire modules QLQ-C30 and BN20 will be used to assess patients' QoL. These internationally recognized and well-validated instruments cover 26 QoL domains. Based on previous studies, particular emphasis will be placed on domains especially relevant to brain tumor patients, including global health status, physical functioning, social functioning, cognitive functioning, communication deficits, and motor dysfunction.
  The questionnaires are designed for completion within approximately 10 minutes, both in the pretreatment phase and during ongoing treatment. Their validity has been demonstrated across various cancer populations and disease stages, including different treatment contexts. Test-retest reliability assessed over a four-day interval has shown good to excellent consistency across all functional domains, with Pearson's r values ranging from 0.72 to 0.91.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schneider M, Potthoff AL, Karpel-Massler G, Schuss P, Siegelin MD, Debatin KM, Duffau H, Vatter H, Herrlinger U, Westhoff MA. The Alcatraz-Strategy: a roadmap to break the connectivity barrier in malignant brain tumours. Mol Oncol. 2024 Dec;18(12):2890-2905. doi: 10.1002/1878-0261.13642. Epub 2024 Apr 3. PMID 38567664
- [Background] Schneider M, Potthoff AL, Ahmadipour Y, Borger V, Clusmann H, Combs SE, Czabanka M, Duhrsen L, Etminan N, Freiman TM, Gerlach R, Gessler F, Giordano FA, Gkika E, Goldbrunner R, Guresir E, Hamou H, Hau P, Ille S, Jagersberg M, Keric N, Khaleghi-Ghadiri M, Konig R, Konczalla J, Krenzlin H, Krieg S, McLean AL, Layer JP, Lehmberg J, Malinova V, Meyer B, Meyer HS, Miller D, Muller O, Musahl C, Pregler BEF, Rashidi A, Ringel F, Roder C, Rossler K, Rohde V, Sandalcioglu IE, Schafer N, Schaub C, Schmidt NO, Schubert GA, Seidel C, Seliger C, Senft C, Shawarba J, Steinbach J, Stocklein V, Stummer W, Sure U, Tabatabai G, Tatagiba M, Thon N, Timmer M, Wach J, Wagner A, Wirtz CR, Zeiler K, Zeyen T, Schuss P, Surges R, Fuhrmann C, Paech D, Schmid M, Borck Y, Pietsch T, Struck R, Radbruch A, Helmstaedter C, Nemeth R, Herrlinger U, Vatter H. The ATLAS/NOA-29 study protocol: a phase III randomized controlled trial of anterior temporal lobectomy versus gross-total resection in newly-diagnosed temporal lobe glioblastoma. BMC Cancer. 2025 Feb 20;25(1):306. doi: 10.1186/s12885-025-13682-3. PMID 39979825
- [Background] Borger V, Hamed M, Ilic I, Potthoff AL, Racz A, Schafer N, Guresir E, Surges R, Herrlinger U, Vatter H, Schneider M, Schuss P. Seizure outcome in temporal glioblastoma surgery: lobectomy as a supratotal resection regime outclasses conventional gross-total resection. J Neurooncol. 2021 Apr;152(2):339-346. doi: 10.1007/s11060-021-03705-x. Epub 2021 Feb 7. PMID 33554293
- [Background] Schneider M, Potthoff AL, Keil VC, Guresir A, Weller J, Borger V, Hamed M, Waha A, Vatter H, Guresir E, Herrlinger U, Schuss P. Surgery for temporal glioblastoma: lobectomy outranks oncosurgical-based gross-total resection. J Neurooncol. 2019 Oct;145(1):143-150. doi: 10.1007/s11060-019-03281-1. Epub 2019 Sep 4. PMID 31485921
- [Background] Karschnia P, Young JS, Dono A, Hani L, Sciortino T, Bruno F, Juenger ST, Teske N, Morshed RA, Haddad AF, Zhang Y, Stoecklein S, Weller M, Vogelbaum MA, Beck J, Tandon N, Hervey-Jumper S, Molinaro AM, Ruda R, Bello L, Schnell O, Esquenazi Y, Ruge MI, Grau SJ, Berger MS, Chang SM, van den Bent M, Tonn JC. Prognostic validation of a new classification system for extent of resection in glioblastoma: A report of the RANO resect group. Neuro Oncol. 2023 May 4;25(5):940-954. doi: 10.1093/neuonc/noac193. PMID 35961053
- [Background] Roh TH, Kang SG, Moon JH, Sung KS, Park HH, Kim SH, Kim EH, Hong CK, Suh CO, Chang JH. Survival benefit of lobectomy over gross-total resection without lobectomy in cases of glioblastoma in the noneloquent area: a retrospective study. J Neurosurg. 2019 Mar 1;132(3):895-901. doi: 10.3171/2018.12.JNS182558. Print 2020 Mar 1. PMID 30835701
- [Background] Schneider M, Ilic I, Potthoff AL, Hamed M, Schafer N, Velten M, Guresir E, Herrlinger U, Borger V, Vatter H, Schuss P. Safety metric profiling in surgery for temporal glioblastoma: lobectomy as a supra-total resection regime preserves perioperative standard quality rates. J Neurooncol. 2020 Sep;149(3):455-461. doi: 10.1007/s11060-020-03629-y. Epub 2020 Sep 29. PMID 32990861
- See also: ATLAS/NOA-29 Website — https://www.ukbonn.de/neurochirurgie/forschung/onkologische-forschung/clinical-trials/atlas-trial/